CLINICAL TRIAL: NCT06873659
Title: A Phase I Dose Escalation and Expansion Study to Evaluate the Safety, Tolerability, Efficacy, Pharmacokinetics, and Pharmacodynamics of SON-DP in Subjects With Advanced Solid Tumors
Brief Title: SON-DP in Participants With Relapsed/Refractory Intolerant to Standard of Care Therapies for Advanced/Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Qurgen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SON-DP-A003-ST
Record Dates: First submitted 2025-03-07; First posted 2025-03-13 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-03

CONDITIONS: Solid Tumor; Gastric Cancer; Liver Cancer
Keywords: SON-DP; Solid Tumor; Gastric Cancer; Liver Cancer
MeSH Terms: conditions — Stomach Neoplasms; Liver Neoplasms

STUDY DESIGN:
Intervention Model Description: Sequential assignment and dose expansion of RP2D in selected tumor types. This is an open-label clinical trial for patients with advanced solid tumors. The design follows an accelerated titration combined with the traditional 3+3 dose escalation rule to ensure the safety of the participants, while also obtaining key information about SON-DP when administering it to subjects who have signed informed consent. In order to minimize the number of participants in dose groups with limited antitumor activity but relatively low toxic side effects. Since the primary objective of this study is to gather information on the antitumor activity of SON-DP and determine the RP2D (Recommended Phase 2 Dose), various methods to assess drug activity have been designed to evaluate the safety, antitumor efficacy, and RP2D of the product.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (8):
- Dose escalation, Cohort 1 (Experimental): SON-DP 3 or 6 participants with solid tumor will be treated with SON-DP by 150-minute IV infusion in the cohort 1 at 2mg/kg dose level once per week in 28-day cycle, for up to 6 cycles.
  Interventions: Drug: SON-DP
- Dose escalation, Cohort 2 (Experimental): SON-DP 3 or 6 participants with solid tumor will be treated with SON-DP by 150-minute IV infusion in the cohort 2 at 3mg/kg dose level once per week in 28-day cycle, for up to 6 cycles.
  Interventions: Drug: SON-DP
- Dose escalation, Cohort 3 (Experimental): SON-DP 3 or 6 participants with solid tumor will be treated with SON-DP by 150-minute IV infusion in the cohort 3 at 4.5mg/kg dose level once per week in 28-day cycle, for up to 6 cycles.
  Interventions: Drug: SON-DP
- Dose escalation, Cohort 4 (Experimental): SON-DP 3 or 6 participants with solid tumor will be treated with SON-DP by 150-minute IV infusion in the cohort 4 at 6mg/kg dose level once per week in 28-day cycle, for up to 6 cycles.
  Interventions: Drug: SON-DP
- Dose escalation, Cohort 5 (Experimental): SON-DP Up to 12 participants with solid tumor will be treated with SON-DP by 150-minute IV infusion at the RP2D-1 dose level once per week for up to 6 cycles.
  Interventions: Drug: SON-DP
- Dose escalation, Cohort 6 (Experimental): SON-DP Up to 12 participants with solid tumor will be treated with SON-DP by 150-minute IV infusion at the RP2D dose level once per week for up to 6 cycles.
  Interventions: Drug: SON-DP
- Dose expansion, Arm 1 (Experimental): SON-DP Up to 24 participants with advanced primary gastric cancer will be treated with SON-DP by 150-minute IV infusion at the RP2D dose level once per week for up to 6 cycles.
  Interventions: Drug: SON-DP
- Dose expansion, Arm 2 (Experimental): SON-DP Up to 24 participants with advanced primary liver cancer will be treated with SON-DP by 1500-minute IV infusion at the RP2D dose level once per week for up to 6 cycles.
  Interventions: Drug: SON-DP

INTERVENTIONS:
Drug: SON-DP — Solution for IV administration

SUMMARY:
A Phase I Dose Escalation and Expansion Study to Evaluate the Safety, Tolerability, Efficacy, Pharmacokinetics, and Pharmacodynamics of SON-DP in Subjects with Advanced Solid Tumors

DETAILED DESCRIPTION:
* SON-DP is different from the conventional cancer cell-killing therapy which have high side effect, drug resistance, cancer recurrence and tumor heterogenicity, SON-DP is a novel transcription factor (TF) protein anticancer drug to treat the Participants with relapsed and advanced metastatic solid tumors. Proposed as an effective therapeutic drug product for a cell-converting cancer therapy, SON-DP is expected to transform cancer cells in situ into normal tissue cells via a SON-DP induced cancer cell reprogramming and re-differentiation process as an innovative rationale.
* SON-DP is developed based on the rationale of cancer cell conversion into normal tissue cells as the primary mechanism of actions of a new cancer therapy, not by cancer cell-killing, the traditional goals of chemotherapy, radiation therapy, targeted therapy and immune therapy. Cancer cell conversion is achieved by the SON-DP induced pluripotent re-programming in situ inside tumor tissue into transient iPSCs (tiPSCs) that quickly re-differentiate into normal tissue cells induced by the differentiating resident tissue environment. The in situ generated tiPSCs either secrete exosomes, providing the embryonic stem cells (ESC)-like microenvironments to transform the surrounding cancer cells into normal tissue cells for an overall malignant phenotype reversion (OMPR) (an effect named as a bystander effect), or display a targeting effect that enables the in situ generated tiPSCs to track down the distant metastatic cancer cells for OMPR (an effect named as a tropism effect). The SON-DP-induced cell reprogramming also restored the mutation-caused and compromised p53 checkpoint in cancer cells to re-establish cell quality control system that ensures the downstream re-differentiation of the in situ generated tiPSCs into normal tissue cells. Overall, this SON-DP-induced re-programming and re-differentiation process is capable of transforming both primary and metastatic cancer cells into normal tissue cells.

  * Preclinical studies demonstrated that treatment of tumors with SON-DP resulted in eradication of late-stage cancers and long term (over 3 years) survival without teratoma formation and cancer recurrence in multiple tumor-bearing mouse/rat (syngeneic) or human xenograft rodent models, providing high treatment efficacy of this cell-converting cancer therapy. Thus, the cell-converting cancer therapy rationale represents a new cancer therapeutic strategy. SON-DP was tolerated in tumor-bearing rodents, as well as in naïve rats, dogs, and monkeys as demonstrated by GLP-enabled (rats and dogs) and non-GLP (monkey) toxicity study and after repeated IV administrations at higher doses compared with the planned clinical dose range. Therefore, the current nonclinical studies, including pharmacodynamics (PD), pharmacokinetics (PK) and toxicology studies, support the safety and efficacy of SON-DP TF protein drug product to be used in clinical studies of human participants. This clinical study will be conducted in selected types of relapsed/refractory advanced/metastatic solid tumors as a step in demonstrating the utility of this anticancer agent.
  * In this SON-DP-A003-ST clinical trial, SON-DP is given to the participants with late stage solid tumors through 150-minutes IV infusion once a week at 4 dose levels during the first Phase I dose escalation to find the recommended phase II dose (RP2D) for the second Phase Ib does expansion stage that will focus on 2 cancer types including advanced primary liver cancer and advanced primary gastric cancer.
  * During Phase Ia dose escalation stage, an 3+3 design will be followed. Phase Ia will enroll the participants with various types of solid tumors that metastasized and not response to standard treatment.
  * During Phase Ib dose expansion stage, SON-DP will be used, at RP2D dose level, to treat the participants with 2 specific cancer types including advanced primary liver cancer and advanced primary gastric cancer. Two groups of cancer cohorts will be opened with eligible participants who have relapsed/refractory/intolerant to standard of care therapies of these two advanced/metastatic solid tumors. Participants will be followed for safety, confirmation of the RP2D, PK, PD, and anti-tumor activity as measured by standard assessment tools.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants aged 18 to 75 years (inclusive).
2. For Phase Ia: Participants with histologic diagnosis and confirmed solid tumor; For Phase Ib: Participants with one of the two tumor types: Group 1: advanced primary liver cancer; Group 2: Advanced primary gastric cancer (including gastroesophageal junction adenocarcinoma).
3. There must be at least one measurable lesion defined by RECIST v1.1. Lesions intended for biopsy should generally not be selected as target lesions, unless the investigator assesses that the biopsy of the lesion will not affect subsequent tumor evaluations. Lesions that have previously undergone radiation therapy, interventional therapy, or other local treatments should generally not be selected as target lesions, unless the lesion shows clear radiological progression after local treatment.
4. The ECOG performance status ≤ 1.
5. Able to understand and willing to sign the informed consent form (ICF) and comply with all the requirements of the protocol.
6. The investigator assesses that the subject's expected lifespan is greater than 3 months.
7. Subjects must be candidates for and agree to the placement of a central venous access line and further must be able, in the opinion of the Investigator, to manage care of this line.
8. Subjects with treated brain metastases are allowed but should be neurologically stable (for 4 weeks post-treatment as assessed by CNS imaging and prior to study enrollment) and off steroids for at least 2 weeks before administration of any study treatment.
9. All subjects in Phase Ia (with partial exceptions for the first 2 dose levels and designated subjects in Phase Ib must be prepared to undergo 2 or more tumor biopsies, one during the screening period and 1-2 biopsy during therapy. In the Investigator's assessment, these biopsies should be feasible considered, safe by the investigator, and not expected to interfere with all other study assessments.
10. Adequate hepatic/renal function as evidenced by meeting all the following requirements:

    1. Total bilirubin ≤ 1.5 × ULN except for subjects with Gilbert's syndrome who are excluded if TBIL > 3.0×ULN or direct bilirubin < 1.5×ULN. And there is no evidence of sustained liver function elevation (within 7 days) or acute hepatic decompensation, as assessed by the investigator.
    2. AST < 3.0×ULN, except for subjects that have tumor involvement of the liver, who are included if AST ≤ 5×ULN. And there is no evidence of sustained liver function elevation (within 7 days) or acute hepatic decompensation, as assessed by the investigator.
    3. ALT ≤ 3.0×ULN, except for subjects that have tumor involvement of the liver, who are included if ALT ≤ 5×ULN. And there is no evidence of sustained liver function elevation (within 7 days) or acute hepatic decompensation, as assessed by the investigator.
    4. Blood Urea Nitrogen (BUN) < 2.5×ULN.
    5. The calculated creatinine clearance (CrCL) using the Cockcroft-Gault formula must be ≥ 60 mL/min.
11. Primary liver cancer: Child-Pugh class A or class B with a score of 7, and no history of hepatic encephalopathy.
12. The subject must have adequate bone marrow function (no blood transfusions or hematopoietic growth factor support within 14 days prior to the first dose of SON-DP), with special circumstances to be jointly evaluated by the study team, sponsor, and CRO medical team:

    1. Absolute neutrophil count (ANC) ≥ 1.5 × 10⁹/L;
    2. Hemoglobin (HGB) ≥ 80 g/L;
    3. Platelet count (PLT) ≥ 75 × 10⁹/L.。
13. Coagulation tests within an acceptable range defined by the following:

    1. Activated partial thromboplastin time (APTT) ≤ 1.5×ULN.
    2. International normalized ratio (INR) or Prothrombin Time (PT) ≤ 1.5×ULN. Exception: INR 2 to ≤ 3 ULN is acceptable for subjects on stable therapeutic anticoagulants without active bleeding within 14 days prior to the first dose of the study drug.
14. Toxicity related to previous antitumor treatments must have returned to baseline or ≤ grade 1 (NCI-CTCAE 5.0), except for toxicities judged by the investigator to pose no safety risk, such as: hair loss, ≤ grade 2 peripheral neuropathy, thyroid dysfunction stabilized by hormone replacement therapy, or other toxicities that are still grade 2 but are assessed by the investigator as chronic, stable, and with no clear safety concerns.
15. Female participants must agree not to breastfeed starting at screening and throughout the study period and for 90 days after final SON-DP administration.
16. Fertile, eligible subjects (both male and female) must agree to use reliable contraception methods (hormonal, barrier methods, or abstinence) during the trial and for at least 90 days after the last dose of the medication.

Exclusion Criteria:

1. Pregnant or breastfeeding women. Pregnancy is defined as the state from conception until the termination of pregnancy, confirmed by a positive human chorionic gonadotropin (hCG) laboratory test. Unless one of the following criteria is met: permanent sterilization (hysterectomy, bilateral salpingectomy, or bilateral oophorectomy), or documented biological or physiological evidence of postmenopausal status (defined as no menstruation for more than 12 months without other conditions), or women who have been menopausal for 6-12 months must have a serum follicle-stimulating hormone (FSH) level > 40 mIU/mL to confirm menopause; otherwise, female subjects will be considered fertile.
2. Participation in an interventional, investigational study within 2 weeks or 5 half-lives, whichever is shorter of the first dose of study treatment.
3. Presence of overt leptomeningeal or active central nervous system (CNS) metastases or primary tumors or CNS metastases that require local CNS-directed therapy (e.g., radiotherapy or surgery) or increasing doses of corticosteroids within the prior 2 weeks.
4. Impaired cardiac function or clinically significant cardiac disease, including any of the following:

   1. Clinically significant and/or uncontrolled heart disease such as congestive heart failure requiring treatment (New York Heart Association [NYHA] Grade ≥ 2), left ventricular ejection fraction (LVEF) < 50% as determined by multiple gated acquisition (MUGA) or echocardiogram (ECHO), uncontrolled hypertension, or clinically significant arrhythmia.
   2. QT interval corrected for heart rate using Fridericia's formula (QTcF) > 470 ms ECG or congenital long QT syndrome at the Screening Visit, except subjects with pacemaker.
   3. Acute myocardial infarction or unstable angina pectoris < 6 months prior to study entry.
5. Uncontrolled hypertension (systolic blood pressure >160 mmHg and diastolic blood pressure >100 mmHg), or in the opinion of the Investigator: a recent history of hypertension crisis, or a recent history of hypertensive encephalopathy.
6. History of stroke or clinically significant intracranial hemorrhage within 6 months before first dose of study drug.
7. Concurrent severe pulmonary diseases, including but not limited to pulmonary embolism within 3 months prior to enrollment, severe asthma, severe chronic obstructive pulmonary disease (COPD), restrictive lung disease, or pneumonia considered based on imaging examination or investigator assessment at screening, as well as a history of non-infectious pneumonia requiring steroid treatment within 12 months prior to signing informed consent.
8. Subject with active human immunodeficiency virus (HIV) infection or a history of HIV infection; subjects with active chronic hepatitis B or active chronic hepatitis C (excluding hepatitis B virus carriers, those with stable hepatitis B after antiviral treatment [HBV DNA negative/ below the lower limit of detection in hospital's quantitative testing or < 500 IU/mL], and HCV-Ab positive but HCV-RNA negative subjects); subject with active syphilis.
9. Other primary malignancies, past or present, except for the enrollment indications of this study. However, this does not include: malignancies that have been cured within 2 years prior to the first dose of SON-DP with no signs of recurrence, fully treated and completely resected cervical carcinoma in situ, completely resected skin basal cell carcinoma or squamous cell carcinoma, any malignancy considered indolent and not requiring treatment, or any type of carcinoma in situ that has been completely resected.
10. The presence of clinically symptomatic, poorly controlled pleural effusion, pericardial effusion, or ascites that requires repeated drainage.
11. Anticancer therapy within 5 half-lives or 3 weeks (whichever is shorter) prior to study entry. Chinese anticancer medicine, three weeks prior first dosing.
12. Received radical radiation therapy or radiation to an area where the bone marrow proportion is greater than 30% within 4 weeks prior to the first dose of SON-DP. Exceptions include: palliative radiation therapy for localized lesions (e.g., radiation therapy for bone lesions aimed at symptom relief) or local interventional treatments (such as transarterial chemoembolization [TACE] and others) assessed by the investigator as posing no safety risks.
13. Subjects receiving systemic chronic steroid therapy or any immunosuppressive therapy (≥ 10 mg/day prednisone or equivalent) two weeks prior first SON-DP dosing. Topical, inhaled, nasal, and ophthalmic steroids are allowed.
14. The use of any live vaccines or live attenuated vaccines against infectious diseases within 4 weeks prior to the first dose of SON-DP and during the study treatment period.
15. Subjects with a history of stroke or having active neurological symptoms, with the exception of chronic conditions or sequelae which in the opinion of the neurologist, Investigator, and the Sponsor, would not impact ongoing neurologic assessments while on study treatment.

    a) This includes subjects with active sickle-cell disease with CNS involvement and active intracranial bleeding.
16. Subjects who are using medications that cannot be used concurrently with urea; subjects who are using medications that require special caution or careful consideration when used with urea. Enrollment may be allowed if the investigator assesses that the risks can be controlled.
17. Subjects with diseases affecting the thirst recognition center, such as central diabetes insipidus, syndrome of inappropriate antidiuretic hormone secretion (SIADH), etc.
18. Active infection requiring intravenous systemic antibiotic or antiviral therapy within 14 days prior to the first dose of SON-DP.
19. Major surgery within 4 weeks of the first dose of study treatment (mediastinoscopy, insertion of a central venous access device, and insertion of a feeding tube are not considered major surgery).
20. Subjects who have undergone solid organ or hematopoietic stem cell transplantation within 5 years prior to signing the informed consent for this study.
21. Any medical condition that would, in the Investigator's judgment, prevent the subject's participation in the clinical study due to safety concerns, compliance with clinical study procedures, or interpretation of study results.
22. Allergy to study protein drug or components of its formulation such as PEI and urea.
23. History of a Grade 3 to 4 allergic reaction to treatment with another protein product.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-02-26 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Number of participants with AEs, with abnormal vital signs, abnormal ECG readings, abnormal clinical laboratory tests results, abnormal physical examinations and abnormal ECOG performance status. | Up to 7 months after the first dose
MTD (Maximum tolerable dose) / RP2D (Recommended dose for phase II) | 28 days post first administration of SON-DP

SECONDARY OUTCOMES:
ORR | Up to 6 months after the first dose. Up to 9 months if treated for 9 cycles.
  Objective response rate (ORR)
DCR | Up to 6 months after the first dose
  Disease control rate (DCR)
TTP | Up to 6 months after the first dose
  Time-to-event endpoints of time to disease progression (TTP)
DOR | Up to 6 months after the first dose
  Duration of response (DoR)
PFS | Up to 6 months after the first dose
  Progression-free survival (PFS)
OS | Up to 12 months after the first dose
  Overall Survival (OS)
Cmax | Up to 6 months after the first dose
  Maximum serum concentration (Cmax) of 3 proteins from SON-DP will be investigated.
Tmax | Up to 6 months after the first dose
  Time to maximum serum concentration (Tmax) of 3 proteins from SON-DP will be investigated.
T1/2 | Up to 6 months after the first dose
  Half-life (T1/2) of 3 proteins from SON-DP will be investigated.
AUC0-t | Up to 6 months after the first dose
  AUC0-t is defined as area under the serum concentration-time curve from time 0 to the time of the last measurable concentration.
CL | Up to 6 months after the first dose
  Clearance (CL) in the serum of 3 proteins from SON-DP per unit of time will be investigated.

OTHER OUTCOMES:
SON-DP concentration in tumor biopsy tissue | Up to 5 weeks after the first dose

CONTACTS AND LOCATIONS:
Locations (10):
- China (10):
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Beijing GoBroad Hospital, Beijing, Beijing Municipality
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Xi 'an Jiaotong University, Xi'an, Shaanxi
  - Introduction to Cancer Hospital of Shandong First Medical University (Shandong Cancer Institute,Shandong Cancer Hospital), Jinan, Shandong
  - ZhongShan Hospital Fudan University, Shanghai, Shanghai Municipality
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No